CLINICAL TRIAL: NCT04974788
Title: Examination of Acute Effects of Different Intensity Respiratory Muscle Training on Respiratory Muscle Activations
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Abant Izzet Baysal University (Other)
Responsible Party: Principal Investigator, Ceyhun Topcuoğlu, Principal Investigator, Abant Izzet Baysal University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AIBU-FTR-CT-03
Record Dates: First submitted 2021-07-09; First posted 2021-07-23 (Actual); Last update posted 2022-10-28 (Actual); Status verified 2022-10

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Chronic Obstructive Pulmonary Disease; Surface EMG; Ventilation; Respiratory Muscle Training
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Respiratory Aspiration

STUDY DESIGN:
Intervention Model Description: Three groups with a conventional therapy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Low Intensity Respiratory Muscle Training Group (Active Comparator): Low intensity respiratory muscle training will be applied to those with chronic obstructive pulmonary disease. Respiratory muscle training will be performed at 30% (low intensity) of the maximum inspiratory pressure, which indicates respiratory muscle strength.
  Interventions: Other: Low Intensity Respiratory Muscle Training
- Medium Intensity Respiratory Muscle Training Group (Active Comparator): Medium intensity respiratory muscle training will be applied to those with chronic obstructive pulmonary disease. Respiratory muscle training will be performed at 60% (medium intensity) of the maximum inspiratory pressure, which indicates respiratory muscle strength.
  Interventions: Other: Medium Intensity Respiratory Muscle Training
- High Intensity Respiratory Muscle Training Group (Active Comparator): High intensity respiratory muscle training will be applied to those with chronic obstructive pulmonary disease. Respiratory muscle training will be performed at 80% (high intensity) of the maximum inspiratory pressure, which indicates respiratory muscle strength.
  Interventions: Other: High Intensity Respiratory Muscle Training

INTERVENTIONS:
Other: Low Intensity Respiratory Muscle Training — Respiratory muscle training will be performed at 30% (low intensity) of the maximum inspiratory pressure, which indicates respiratory muscle strength. The training will consist of 2 sessions in total; Each session will last 15 minutes. There will be a break of at least 30 minutes between training sessions.
  Arms: Low Intensity Respiratory Muscle Training Group
Other: Medium Intensity Respiratory Muscle Training — Respiratory muscle training will be performed at 60% (medium intensity) of the maximum inspiratory pressure, which indicates respiratory muscle strength. The training will consist of 2 sessions in total; Each session will last 15 minutes. There will be a break of at least 30 minutes between training sessions.
  Arms: Medium Intensity Respiratory Muscle Training Group
Other: High Intensity Respiratory Muscle Training — Respiratory muscle training will be performed at 80% (high intensity) of the maximum inspiratory pressure, which indicates respiratory muscle strength. The training will consist of 2 sessions in total; Each session will last 15 minutes. There will be a break of at least 30 minutes between training sessions.
  Arms: High Intensity Respiratory Muscle Training Group

SUMMARY:
It has been observed in the literature that respiratory muscle electromyography activations at certain threshold loads have been examined in individuals with chronic obstructive pulmonary disease. However, no study has been found in the literature examining the acute effects of respiratory muscle training given at low, medium and high threshold loads on respiratory muscle activations. With this planned study, it is aimed to examine the electromyography activations of respiratory muscles before and after respiratory muscle training and to contribute to the literature by comparing the acute effects of respiratory muscle training applied at low, medium and high intensity on respiratory muscle electromyography activations.

DETAILED DESCRIPTION:
Chronic obstructive pulmonary disease is a common, preventable and treatable disease characterized by persistent respiratory symptoms and airway limitation due to airway and/or alveolar abnormality, which is affected by many factors that cause abnormal lung development resulting from exposure to harmful gases or particles. Chronic obstructive pulmonary disease is known as the fourth most common cause of death in the world and is expected to rise to third place by the end of 2020. Physiopathological changes such as airflow limitation, bronchial fibrosis, increased airway resistance, ciliary dysfunction, gas exchange abnormalities and air trapping occur in Chronic obstructive pulmonary disease. While smoking is the most common risk factor in chronic obstructive pulmonary disease; Occupational dust and chemicals, air pollution, lung growth and development, genetic predisposition such as age and gender, and exposure to environmental effects. Symptoms such as shortness of breath (dyspnea), cough and sputum are common in chronic obstructive pulmonary disease. In addition to pulmonary changes such as increased respiratory workload, there are also extrapulmonary changes such as respiratory muscle dysfunction in individuals with chronic obstructive pulmonary disease.

Respiratory muscle dysfunction; It is a decrease in respiratory muscle strength, endurance, or both, caused by factors such as elongated diaphragm fibers, increased respiratory workload, changes in muscle mass and abdominal weight. Strength is defined as the muscle's capacity to produce power, while endurance is defined as the muscle's ability to sustain a given force over time (the capacity to resist fatigue). Loss of strength and/or endurance contributes to diaphragm weakness and impaired performance.

Neural respiratory impulse, indirectly measured by electromyogram of respiratory muscles, has attracted attention as a potential physiological marker of clinical deterioration due to imbalance between workload and capacity of respiratory muscles. The neural respiratory drive is the output of the brainstem respiratory centers. Neural respiratory drive is not affected by the patient's will, is associated with symptoms such as dyspnea, and is usually increased in chronic obstructive pulmonary disease patients.

Mechanical abnormalities such as airflow obstruction, static and dynamic hyperinflation, and intrinsic positive end-expiratory pressure increase the load on respiratory muscles in individuals with chronic obstructive pulmonary disease. Inspiratory muscle contraction is impaired as a result of pressure changes, muscle shortening, increased contraction rate, change in geometry, and decreased compliance of the respiratory system. As a result, an increase in muscle activation and neural respiratory drive is observed. Those with severe chronic obstructive pulmonary disease require significantly higher muscle activations, both electrical and mechanical, to breathe and overcome the respiratory workload than those with mild to moderate chronic obstructive pulmonary disease. In individuals with chronic obstructive pulmonary disease, neural respiratory drive increases when the load on the respiratory muscles increases as a result of an increase in respiratory workload, a decrease in capacity, or a combination of both. Studies have shown that in addition to respiratory workload, workloads given with respiratory muscle training devices lead to an increase in the activation of respiratory muscles.

In addition to pulmonary changes, extrapulmonary changes occur in individuals with chronic obstructive pulmonary disease. Loss of respiratory muscle strength and endurance; The effect of the inappropriate position of the diaphragm on length-tension due to hyperinflation are among the most common extrapulmonary changes resulting from the use of corticosteroids, hypoxemia and hypercapnia. Weakness of respiratory muscles in chronic obstructive pulmonary disease patients leads to hypoxemia, hypercapnia, dyspnea and reduces exercise capacity. Inspiratory muscle training reduces type 2 fibers, shortens the inspiratory time, prolongs the expiratory time, and reduces dynamic hyperinflation. Inspiratory muscle training has been proposed as one of the non-pharmacological treatment modalities because it can delay worsening of lung function by increasing inspiratory muscle strength and endurance. In chronic obstructive pulmonary disease, inspiratory muscle training improves respiratory muscle strength and exercise capacity and reduces dyspnea and is widely used in therapy.

ELIGIBILITY:
Inclusion Criteria:

* Individuals diagnosed with chronic obstructive pulmonary disease
* Be between the ages of 40-75
* No medication changes due to acute exacerbation for at least three weeks
* Be stable
* Volunteering to participate in research
* To cooperate
* Patients with written consent form
* Healthy individuals in a similar age range without a diagnosed disease and symptoms will be included

Exclusion Criteria:

* Those with a history of chronic obstructive pulmonary disease exacerbations
* Individuals with orthopedic disease
* Individuals with neurological disease
* Individuals with other co-existing lung and systemic diseases other than chronic obstructive pulmonary disease
* Those who have had major surgery in the past few months
* Individuals with a history of recurrent significant clinical infections
* Have cognitive problems
* Having had unstable angina,
* Previous Myocardial Infarction
* Individuals with severe congestive heart failure refractory to medical therapy, individuals with uncontrolled hypertension
* Individuals with cancer

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-06-30 (Estimated); Primary Completion 2023-07-30 (Estimated); Study Completion 2023-08-30 (Estimated)

PRIMARY OUTCOMES:
Surface Electromyography (EMG) | 45 minutes
  Activation of respiratory muscles will be performed with a surface Electromyography (EMG) device. The measurement will be performed by placing Electromyography (EMG) electrodes on the motor points of the respiratory muscles. Increased respiratory muscle activations indicate that respiratory muscles are used more; The decrease in respiratory muscle activations indicates that the respiratory muscles are used less.

SECONDARY OUTCOMES:
Pulmonary Function Test | 10 minutes
  Pulmonary function test will be performed with a spirometer according to the criteria of the American Thoracic Society (ATS) and the European Respiratory Society. While the decrease in pulmonary function test parameters shows worsening of lung functions; parameters in the normal range indicate good lung functions.
Measurement of Maximal Inspiratory Pressure | 5 minutes
  Maximal Inspiratory Pressure will be measured with an intraoral pressure measuring device. Maximal Inspiratory Pressure reflects respiratory muscle strength. An increase in Maximal Inspiratory Pressure indicates high respiratory muscle strength; A low Maximal Inspiratory Pressure value indicates respiratory muscle weakness.
Chronic Obstructive Pulmonary Disease Assessment Test (CAT): | 5 minutes
  Chronic Obstructive Pulmonary Disease Assessment Test is an eight-item scale measuring health status in Chronic Obstructive Pulmonary Disease. This scale is used to determine the health status of individuals with Chronic Obstructive Pulmonary Disease all over the world. Each question is scored between 0-5 and a total score between 0 and 40 is given. A score of 0 represents the best and a score of 40 represents the worst state of health.
Modified Medical Research Council Dyspnea Scale: | 2 minutes
  It is a 5-item scale scored between 0-4 for individuals' shortness of breath. Evaluates dyspnea and activity limitation in individuals with chronic obstructive pulmonary disease. An increase in the score indicates an increase in shortness of breath.
Modified Borg Scale (MBS): | 2 minutes
  In this scale, in which the perception of shortness of breath at rest and during exercise will be evaluated, scoring varies between 0-10 points, although high scores indicate high breathlessness and fatigue.

IPD SHARING:
Plan to Share IPD: No